CLINICAL TRIAL: NCT01513863
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Design, Multi-Site Clinical Study to Compare the Bioequivalence of Two Metronidazole 1% Topical Gel Formulations in Patients With Moderate to Severe Rosacea
Brief Title: A Therapeutic Equivalence Study of Two Metronidazole 1%Topical Gel Treatments for Patients With Rosacea
Acronym: MTZG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTZG 1101
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metronidazole Topical Gel 1% (Experimental)
  Interventions: Drug: Metronidazole Topical Gel 1%
- Metronidazole Topical Gel 1% (Metrogel ) (Active Comparator)
  Interventions: Drug: Metronidazole Topical Gel 1% (Metrogel)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole Topical Gel 1% — Metronidazole Topical Gel 1% applied to affected area once a day for 70 days
  Arms: Metronidazole Topical Gel 1%
Drug: Metronidazole Topical Gel 1% (Metrogel) — Metronidazole Topical Gel 1% applied to affected area once a day for 70 days
  Arms: Metronidazole Topical Gel 1% (Metrogel )
Drug: Placebo — Placebo applied to affected area once a day for 70 days
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate that metronidazole 1% topical gel is effective for the treatment of patients with moderate to severe rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, 18 years of age or older.
2. Signed informed consent form, which meets all criteria of current FDA regulations.
3. If female and of child bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom, IUD, oral, transdermal, injected or implanted hormonal contraceptives).
4. Have moderate to severe facial rosacea.
5. Have a Baseline Investigator Global Evaluation Score of 3 or 4.

Exclusion Criteria:

1. Mild facial rosacea (less than 8 inflammatory lesions on the face) or very severe rosacea (more than 50 inflammatory lesions)
2. Patients with excessive facial hair (beards, sideburns, moustaches, etc.) that would interfere with the diagnosis or assessment of rosacea.
3. History of hypersensitivity or allergy to Metronidazole, or other ingredients of the formulation.
4. Use of oral retinoids (e.g. Accutane ®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed) within the 6 months prior to the baseline visit.
5. Use of the following within 1 month prior to the baseline visit:

   * Topical Retinoids to the face
   * Systemic antibiotics known to have an impact on the severity of facial Rosacea
   * Systemic Steroids
6. The use of anticoagulant therapy within 14 days prior to baseline.
7. The use of any antipruritics, including antihistamines within 24 hours of any study visits.
8. History of blood dyscrasia.
9. Ocular rosacea (e.g., conjunctivitis, blepharitis, keratitis) of sufficient severity to require topical or systemic antibiotics.
10. Any dermatological condition other than rosacea that in the Investigator's opinion may interfere with the evaluation of the Patient's rosacea (e.g., acne, psoriasis, dermatitis).
11. Females who are pregnant, lactating or likely to become pregnant during the study.
12. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study Patient at undue risk by participation.
13. Any Patient (male or female) who has started, or changed hormonal therapy within 3 months of the Baseline visit (this includes hormonal contraceptives).
14. Use of high strength (20% or above) alpha-hydroxy acid for facial peel or any type of chemical facial skin peel or other significant cosmetic procedures within 2 months of the study start.
15. Receipt of any drug as part of a research study within 30 days prior to dosing.
16. Employees of the research center or Investigator.
17. Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Clinical Success | Day 70
  A patient is considered a clinical success if the IGE is 0 (Clear)or 1 (Almost Clear)
Treatment Success | Day 70
  A patient is considered a treatment success if the mean percent change from baseline at week 10 (Day 70) in the inflammatory (papules and pastales) lesion count of Rosacea

SECONDARY OUTCOMES:
Change in Investigational Global Evaluation (IGE) | Day 70
  Mean change from baseline to end of treatment in IGE

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Investigator Site, Phoenix, Arizona
  - Investigator Site, Long Beach, California
  - Investigator Site, Newport Beach, California
  - Investigator Site, Denver, Colorado
  - Investigator Site, Jacksonville, Florida
  - Investigator Site, Miami, Florida
  - Investigator Site, Miramar, Florida
  - Investigator Site, Arlington Heights, Illinois
  - Investigator Site, Plainfield, Indiana
  - Investigator Site, Henderson, Nevada
  - Investigator Site, Hickory, North Carolina
  - Investigator Site, High Point, North Carolina
  - Investigator Site, Wilmington, North Carolina
  - Investigator Site, South Euclid, Ohio
  - Investigator Site, Hazleton, Pennsylvania
  - Investigator Site, Simpsonville, South Carolina
  - Investigator Site, Kingsport, Tennessee
  - Investigator Site, Knoxville, Tennessee
  - Investigator Site, Nashville, Tennessee
  - Investigator Site, San Antonio, Texas
  - Investigator Site, Webster, Texas
  - Investigator Site, West Jordan, Utah